CLINICAL TRIAL: NCT03476772
Title: Nalbuphine as an Adjuvant to Caudal Bupivacaine for Postoperative Analgesia in Children Undergoing Hypospadius Repair
Brief Title: Nalbuphine Plus Caudal Bupivacaine in Hypospadius Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, TKSayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NBCH
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (No Intervention): children undergoing hypospadius repair given 1 ml/kg of bupivicaine 0.25 % via caudal route to achieve post operative analgesia
- B (Active Comparator): children undergoing hypospadius repair given 1 ml/kg of bupivicaine 0.25 % plus 0.1 mg nalbuphine via caudal route to achieve post operative analgesia
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — Children will be randomly assigned into 2 groups of 30 patients each. They will receive caudal anesthesia using bupivacaine 0.25% 1ml/kg plus 2 ml normal saline in the control group, bupivacaine 0.25% 1ml/kg plus nalbuphine 0.1 mg/kg in 2 ml solution in the nalbuphine group.
  Arms: B

SUMMARY:
Caudal aneasthesia for pediatric surgery was first reported in 1933. Since then, studies have described the indications for pediatric caudal block, the level of analgesia, doses, advantages and disadvantages of this technique.

In children, caudal anesthesia is most effectively used as adjunct to general aneasthesia and has an opioid-sparing effect, permitting faster and smoother emergence from aneasthesia.

A single shot caudal anesthesia provides relatively brief analgesia for 4 to 8 hours depending on the agent used. Prolongation of anesthesia can be achieved by adding various adjuvants, such as opioids and nonopioids such as clonidine, ketamine, midazolam, and neostigmine,with varying degrees of success.

DETAILED DESCRIPTION:
The somatic innervation of the lower urogenital system arises principally from the spinal nerves sacral 2 to sacral 4 by way of the pudendal nerve. After passing under the sacrospinous ligament and over the sacrotuberous ligament through Alcock's canal, the pudendal nerve passes through the transverse perineal muscle to course on the dorsum of the penis as the dorsal nerve of the penis. The dorsal nerve of the penis is thought to be a sensory nerve. The autonomic innervation of the penis arises from the vesical and prostatic plexus, which is composed of sympathetic nerves from lumbar 1 and lumbar 2, and parasympathetic nerves from sacral 2 to sacral 4. The cavernosal nerve leaves the pelvis between the transverse perineal muscles and the membranous urethra before passing beneath the arch of pubis to supply each corporal body.

After the pudendal nerve leaves the pudendal canal, two main terminal branches arise, the inferior rectal and the perineal nerves. The function of the inferior rectal nerve is motor innervation of external anal sphincter and is thought to be devoid of urogenital function. Sensory portions of the inferior rectal nerve are important for perianal skin sensation. The perineal nerve has both a motor and sensory component. The motor efferents are known to innervate the pelvic musculature, mainly the bulbospongiosus muscle. To achieve complete anesthesia (analgesia) for hypospadius repair, afferent blockade must be complete at lumbar 1 through sacral 4.

Nalbuphine is a mixed k-agonist and µ-antagonist opioid of the phenanthrene group; it is related chemically to naloxone and oxymorphone. Nalbuphine leads to activation of spinal and supraspinal opioid receptors which leads to good analgesia with minimal sedation, minimal nausea and vomiting, less respiratory depression and stable cardiovascular functions. Safety and efficacy of nalbuphine have been established in the clinical field and its safety and efficacy also established via the epidural route. Nalbuphine was also added in epidural analgesia for adults and provided an increase in the efficacy and the duration of postoperative analgesia. The effect of nalbuphine addition in caudal anesthesia in pediatrics is not well established.

ELIGIBILITY:
Inclusion Criteria:

* Male children undergoing hypospadius repair, with an American Society of Anesthesiologists (ASA) physical status I.

Exclusion Criteria:

* Guardians refusal.
* Contraindication to caudal block such as:

  * Patients with congenital anomalies at the lower spine or meninges.
  * Patients with increased intracranial pressure.
  * Patients with skin infection at the site of injection.
  * Patients with bleeding diathesis.
  * Know allergy to any drug used in this study.

Ages: 2 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
post operative pain measurement | 24 hours
  Postoperative pain intensity Measured by Face, Legs, Activity, Cry & consolability (FLACC) pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SPIEGEL P. Caudal anesthesia in pediatric surgery: a preliminary report. Anesth Analg. 1962 Mar-Apr;41:218-21. No abstract available. PMID 13915759
- [Background] de Beer DA, Thomas ML. Caudal additives in children--solutions or problems? Br J Anaesth. 2003 Apr;90(4):487-98. doi: 10.1093/bja/aeg064. No abstract available. PMID 12644422
- [Background] Lake CL, Duckworth EN, DiFazio CA, Durbin CG, Magruder MR. Cardiovascular effects of nalbuphine in patients with coronary or valvular heart disease. Anesthesiology. 1982 Dec;57(6):498-503. doi: 10.1097/00000542-198212000-00012. PMID 6983316